CLINICAL TRIAL: NCT07117500
Title: Research on the Development and Implementation of an Exercise Rehabilitation Program for Aortic Dissection Patients After Percutaneous Intervention Based on the Behavior Change Wheel Theory
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shuzhen Wang (Other)
Responsible Party: Sponsor-Investigator, Shuzhen Wang, Nurse Practitioner (NP), Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT-I-2025-083
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCW Rehabilitation (Experimental)
  Interventions: Behavioral: Routine; Behavioral: BCW
- Routine Care (Active Comparator)
  Interventions: Behavioral: Routine

INTERVENTIONS:
Behavioral: Routine — Inpatient Care: Continuously monitor vital signs (BP, HR, SpO₂), neurological status, and limb function; administer prescribed antihypertensives with thorough medication education and efficacy tracking. Strictly prohibit Valsalva maneuvers . Assess pain levels, wounds, and psychological state; deliver scheduled analgesics and emotional counseling to maintain stable mood. Implement lifestyle optimization: 7+hr sleep/night, portion-controlled nutrition, and gradual postoperative mobilization.
  Discharge & Follow-up: Enforce BP control through medication adherence. Ban vigorous activities (mountaineering/swimming/competitive sports); allow low-stress aerobics . Distribute Exercise Diaries (Appx 6) mandating daily logs with critical warnings: STOP immediately if nausea, chest pressure, dizziness, dyspnea, or arrhythmia occur and urgent revisit. Require complete tobacco cessation and secondhand smoke avoidance.
Behavioral: BCW — 1.1 Assessment of physical fitness and formulation of individualized exercise rehabilitation plans 1.2 Inpatient Phase (Postoperative Day 1 - Week 1): Monitor via ICU Mobility Scale (IMS) before each session:▪ Score 0 : Passive range of motion (PROM) exercises▪ Scores 1-3 : Active bed-based joint mobility training▪ Scores 4-6 : Standing balance training▪ Scores 7-10 : Ambulatory walking training 1.3 Early Outpatient Phase (Weeks 2-4): Initiate when IMS=10:▪ Perform 6-Minute Walk Test (6MWT) ▪ If distance >450m: Prescribe low-intensity aerobic walking " Speed: 3 km/h" Progression: Start at 10 min/day (≈500 steps), increase by 10 min every other day up to 40 min/day 1.4 Intermediate Rehabilitation (Weeks 5-12): Moderate-intensity aerobic walking + Resistance training :▪ Walking: 4-6 km/h, 30 min/session, 3 sessions/week▪ Resistance training: Seated elastic band exercises, 20 min/session, 2 sessions/week
  Arms: BCW Rehabilitation

SUMMARY:
Study Title ： Effectiveness of a BCW Theory-Based Exercise Rehabilitation Program in Post-Endovascular Aortic Dissection Patients: A Randomized Controlled Trial

Primary Objective ： To determine whether an exercise rehabilitation program constructed based on the Behavior Change Wheel (BCW) framework improves postoperative quality of life (QoL) in patients undergoing endovascular aortic repair (EVAR).

Methodology ： Intervention Group (n= 40): Receives the BCW-based exercise rehabilitation protocol.

Control Group (n= 40): Receives routine care and health education . Outcome Measures ：

Primary Endpoint :QoL changes assessed via validated scales ( SF-36) at:

Pre-discharge (T0)

1 month postoperatively (T1) 3 months postoperatively (T2)

Secondary Endpoints (Daily Monitoring):

Exercise duration (minutes/day) Exercise intensity Post-exercise blood pressure (mmHg) Post-exercise heart rate (bpm)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed aortic dissection diagnosis by CTA and MRI, undergoing endovascular interventions : Thoracic Endovascular Aortic Repair (TEVAR), fenestrated endografting, or branched stent-graft techniques.
2. Conscious and capable of voluntary participation in this study (with documented informed consent).

Exclusion Criteria:

1. Severe concomitant organ diseases, such as coronary artery disease (CAD) , valvular heart disease , ventricular aneurysm , or life-threatening arrhythmias .
2. Patients with unstable angina or myocardial infarction within the past 1 month .
3. Patients with comorbid psychiatric disorders.
4. Patients with active infections or malignant tumors.
5. Presence of pacemakers or implantable cardioverter-defibrillators (ICDs) .
6. Translation : Hemodynamic instability with thrombosis , malperfusion , or coagulopathies.
7. Concurrent participation in other clinical trials .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
SF-36 | Preoperative，1 month postoperative，3 month postoperative

SECONDARY OUTCOMES:
HADS | Preoperative，1 month postoperative，3 month postoperative
  Hospital Anxiety and Depression Scale，HADS
PISQ | Preoperative，1 month postoperative，3 month postoperative
  Pittsburgh Sleep Quality Index
Self-Efficacy for Exercise Scale | Preoperative，1 month postoperative，3 month postoperative
  SEE-C
complications | Within 3 months postoperatively
6MWT | Predischarge ,1 month postoperative，3 month postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided